CLINICAL TRIAL: NCT05778903
Title: Maxillary Nerve Blocks in Children - An MRI Study of the Suprazygomatic
Brief Title: Maxillary Nerve Blocks in Children - An MRI Study of the Suprazygomatic Approach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Axel R. Sauter, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 563605
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Nerve Block; Cleft Palate; Analgesia
MeSH Terms: conditions — Cleft Palate; Agnosia | interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound guided Suprazygomatic Maxillary Nerve Block (Active Comparator): An ultasound guided SMNB is admitted on one half of the patients face (left or right) according to randomiced allocation. 0.15 ml/kg of bupivacaine 0.25 mg/ml with epinephrin 5 mcg/ml is injected.
  Interventions: Other: Nerve block
- Landmark guided Suprazygomatic Maxillary Nerve Block landmark (Active Comparator): A langmark guided SMNB is admitted on the other half of the patients face (left or right) according to randomiced allocation. 0.15 ml/kg of bupivacaine 0.25 mg/ml with epinephrin 5 mcg/ml is injected.
  Interventions: Other: Nerve block

INTERVENTIONS:
Other: Nerve block — Suprazygomatic maxillary nerve block

SUMMARY:
Ultrasound-guided suprazygomatic maxillary nerve block (SMNB) will be performed in paediatric patients with or without the aid of ultrasound guidance. Magnetic resonance imaging (MRI) is used to visualize the spread of the local anaesthetic (LA) spread after suprazygomatic injection and to verify LA contact with the maxillary nerve in the pterygopalatine fossa (PPF).

ELIGIBILITY:
Inclusion Criteria:

* Paediatric patients scheduled for cleft palate (CP) surgery with SMNB as part of their perioperative pain treatment
* American Society of Anesthesiologists physical status 1 - 2
* Age 10 to 24 months
* Given informed written consent by legal guardian

Exclusion Criteria:

* American Society of Anesthesiologists physical status > 2
* Patients with cranial deformation
* Patients with concomitant medical treatments or medical conditions interfering with peripheral nerve block treatment
* Patients with concomitant medical treatments or medical conditions interfering with MRI
* Patients that are allergic to bupivacaine or other local anaesthetic agents.

Ages: 10 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of LA spread into the PPF | day one - within an hour after intervention (peripheral nerve block)
  Local anesthetic spread to the maxillaris nerve in the pterygopalatine fossa detected by MRI (binary outcome)

SECONDARY OUTCOMES:
Rate of LA spread to other anatomical areas and structures | day one - within an hour after intervention (peripheral nerve block)
  Local anaesthetic spread to orbita, nasal cavity, cranial fossa, infratemporal fossa, or other structures detected by MRI (binary outcome)
Rate of hematoma | day one - within an hour after intervention (peripheral nerve block)
  Accumulation of blood detected by MRI (binary outcome)
Superior-inferior needle angle | day one - immediately after intervention (peripheral nerve block)
  Angle of the injection needle meassured in a coronal plane
Anterior-posterior needle angle | day one - immediately after intervention (peripheral nerve block)
  Angle of the injection needle meassured in a sagittal plane
Needle depth | day one - immediately after intervention (peripheral nerve block)
  Depth of the injection needle
Side effects and adverse events | day one
  All side effects or adverse events that might be detected
Postoperative analgesic consumption | day one and day two
  Opioid consumption during the first 24 hours after surgery
MRI time | day one
  Time consumption for MRI

CONTACTS AND LOCATIONS:
Overall Officials: Axel Sauter, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Suleiman NN, Lien I, Akhavi MS, Impieri D, Ullensvang K, Moen JM, Lindholm P, Langesaeter E, Sauter AR. Ultrasound guidance does not improve local anesthetic distribution in suprazygomatic maxillary nerve blocks in pediatric patients: a clinical, randomized, controlled, observer-blinded, crossover MRI trial. Reg Anesth Pain Med. 2025 Apr 11:rapm-2025-106439. doi: 10.1136/rapm-2025-106439. Online ahead of print. PMID 40216530